CLINICAL TRIAL: NCT07075588
Title: Integrating Free-choice Marketplace, dieTitian coacHing, cultuRally Tailored messagIng to improVE Blood Pressure
Acronym: iTHRIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00457380; 25CDA1453103 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-07-17; First posted 2025-07-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Hypertension Complicated With Type 2 Diabetes
Keywords: Digital Farmacy; DASH Diet; Personalized dietitian coaching
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTHRIVE intervention arm (Experimental): iTHRIVE intervention will include access to a digital produce prescription platform, virtual dietitian coaching, a Home blood pressure monitor with App integration, and produce
  Interventions: Behavioral: iTHRIVE intervention
- Comparator Arm (Active Comparator): The active comparator arm will receive enhanced usual care, standard produce bags, general dietary advice, and a home blood pressure monitor
  Interventions: Behavioral: Active comparator

INTERVENTIONS:
Behavioral: iTHRIVE intervention — Integration of three traditionally siloed components:
  1. Digitally enabled food access
  2. Personalized nutrition support
  3. Clinical care-rision of home blood pressure device with app
  Arms: iTHRIVE intervention arm
Behavioral: Active comparator — Active comparator arm will receive enhanced usual care that consists of:
  1. Standard produce bag
  2. Home blood pressure Device without app
  3. General dietary advice
  Arms: Comparator Arm

SUMMARY:
iTHRIVE intervention is a 2-arm randomized controlled trial testing the effects of digital FARMacy, personalized dietitian coaching with produce prescriptions, and home blood pressure measurement in 100 hypertensive adults living in high food priority areas in counties in Maryland.

DETAILED DESCRIPTION:
Cardiovascular-kidney-metabolic (CKM) syndrome is a devastating public health crisis that affects nearly 90% of US adults. CKM accounts for >30% of all US deaths and >5 million hospitalizations annually and imposes an annual economic burden of ≥$1 trillion, with a disproportionate impact on Black, Hispanic adults. Inequitable access to care, high-quality food, culturally tailored dietitian support, and living in "food deserts" (also known as Healthy Food Priority Areas (HFPAs) exacerbate CKM disparities. Innovative approaches are urgently needed to sustainably improve food access and CKM health of Black and Hispanic adults.

More than three times as many Black adults (31%) in Baltimore City live in HFPAs compared to White adults (9%). About 45% of households in Montgomery County earn less than the self-sufficiency standard, 64% of Supplemental Nutrition Assistance Program (SNAP)-eligible adults are unenrolled, the highest rate in MD. In 2022, 48% of Prince George's County residents lived in HFPAs. Reasons for these disparities are complex and comprise factors at the individual, provider, community, and systemic levels.

Evidence-based interventions that improve CKM health include personalized dietitian coaching, home blood pressure monitoring (HBPM), and culturally tailored messages. Digital interventions could improve access to dietitians and fruits/vegetables (f/v) through digital "FARMacy" (akin to a virtual farmers market). Implementation strategies for the delivery of these digital interventions are critical gaps, and clinic integration remains unclear. Digital FARMacy platforms offer potential for increased reach and engagement-relative effectiveness and implementation approach have not been explored.

The investigators propose to test the effects of iTHRIVE using a randomized controlled trial among 100 adult participants living in HFPAs in MD counties with uncontrolled BP defined as systolic blood pressure (SBP) ≥130 milimiters of mercury (mmHg) and diabetes or moderate risk chronic renal disease. Participants will be randomized to either iTHRIVE (digital FARMacy, personalized dietitian coaching with produce prescription [PRx], and HBPM) or enhanced usual care (EUC, general dietary advice, standard food bags). The investigators will assess the effectiveness of iTHRIVE in improving systolic blood pressure at 6 months and evaluate the reach, adoption, implementation, maintenance, and budget impact of iTHRIVE

ELIGIBILITY:
Inclusion Criteria:

* 21-70 years
* Self-identify as Black/African American or Hispanic/Latino
* Have Stage 2 CKM defined as:
* Systolic BP ≥130mmHg (measured at screening) AND at least one of:
* Hypertension (ICD-10: I10-I16)
* Prediabetes (HbA1c 5.7-6.4%) or Type 2 Diabetes (HbA1c ≥6.5%)
* Stage 3 chronic kidney disease (CKD) (eGFR 30-59 mL/min/1.73m²)
* Live in census tracts identified by the Montgomery/ Prince George's/Baltimore City County Departments of Planning as HFPA:
* Healthy Food Availability Index score is low (0-9.5),
* Median household income ≤185% of Federal Poverty Level

  * 30% of households have no vehicle,
* Distance to supermarket >1/4 mile. 5. Have refrigeration, food preparation appliances (microwave, stove), and cell phones for the App

Exclusion Criteria:

* Age <21 years
* Diagnosis of end-stage renal disease (ESRD), dialysis
* Serious medical condition that either limits life expectancy or requires active management (e.g., cancer)
* Significant food allergies, preferences, intolerances, or dietary requirements that would interfere with diet adherence
* Active alcohol or substance use disorder (i.e., not sober/abstinent for ≥ 30 days)
* Patients with cognitive impairment or other condition preventing their participation in the intervention
* Pregnant, breastfeeding, or planning pregnancy
* Current participation in a care management program related to health conditions (e.g., weight reduction, smoking cessation) or another clinical trial that could interfere with the study protocol
* Planning to move out of the geographic area in 12 months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) | Baseline, 3, 6 and 12 months
  Systolic blood pressure measured in millimeters of mercury (mmHg) by the home blood pressure device and in the electronic medical record (EMR)

SECONDARY OUTCOMES:
Hemoglobin A1c (percent) | Baseline, 3, and 6 months
  Hemoglobin A1c
Weight in pounds | Baseline, 3, 6, and 12 months
  Weight will be measured in pounds
Change in Dietary Patterns assessed by 24 hour dietary recall | Baseline and 6 months
  Change in Dietary Approaches to Stop Hypertension (DASH) adherence scores are summarized from 24-hour dietary recall administered by the investigator. Score range 0-9, higher scores indicate better adherence.
Cost effectiveness | Baseline and 12 weeks
  Intervention cost/person will be estimated based on the total cost of the intervention and the estimated cost of treatment
Cultural appropriateness and acceptability assessed by Cultural Sensitivity Assessment Tool | Baseline, 6 and 12 months
  Self-reported acceptance of Data Apps using Cultural Sensitivity Assessment Tool ( CSAT) with a score range of 1 to 4. A score of 2.5 is the cut-off score for acceptability
Height in inches | Baseline, 3,6 and 12months
  Height will be measured in inches

CONTACTS AND LOCATIONS:
Overall Officials: Oluwabunmi Ogungbe, PhD, MPH, RN, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No